CLINICAL TRIAL: NCT03544385
Title: Effect of Ocular Hygiene on Scleral Lens Wear
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Houston (Other)
Responsible Party: Principal Investigator, Amy B. Conner, Resident, Optometry, University of Houston
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: STUDY00000851
Record Dates: First submitted 2018-05-21; First posted 2018-06-01 (Actual); Last update posted 2018-06-01 (Actual); Status verified 2018-05

CONDITIONS: Scleral Contact Lenses
MeSH Terms: interventions — Ringer's Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Group (Experimental)
  Interventions: Drug: Ringers Solution
- Placebo Group (Placebo Comparator)
  Interventions: Drug: Placebo - Concentrate

INTERVENTIONS:
Drug: Ringers Solution — Treatment vs Placebo
  Arms: Treatment Group
Drug: Placebo - Concentrate — treatment vs placebo
  Arms: Placebo Group

SUMMARY:
This is a study to evaluate the performance of Lid Scrubs when added to the daily regimen of scleral lens wear. Lid Scrubs contain surfactants and chemically developed Ringer's solution with microbial attributes. Lid Scrubs are typically used in the treatment of blepharitis. This study is geared towards showing added benefits to scleral lens patients when adding Lid Scrubs to their daily regimens. This study will also show if Lid Scrubs are capable of antimicrobial properties on scleral lens accessories.

ELIGIBILITY:
Inclusion Criteria:

* • Age: 18 years old to - 85 years old Scleral Lens Correction criteria: Patients should be habitual scleral lens wearers. Patients should use scleral lenses for at least 8 hours a day and for at least 5 days of the week

Exclusion Criteria:

* Exclusions to participate in the study include: adults unable to consent, age restrictions, pregnant women, prisoners, non-english speaking patients (as consent forms are only available in the English language), current optometry students and faculty as these patients may be biased to which products they are using.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2018-05-18 (Actual); Primary Completion 2018-07-25 (Estimated); Study Completion 2018-10-25 (Estimated)

PRIMARY OUTCOMES:
length of scleral lens wear | one month

CONTACTS AND LOCATIONS:
Locations (1):
- University of Houston- College of Optometry, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No